CLINICAL TRIAL: NCT06826781
Title: Evaluating Q-Collar Effects on Cerebrovascular Control in Response to Exercise
Brief Title: Evaluating Q-Collar Effects on Brain Blood Flow Control During Exercise
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Spaulding Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, J. Andrew Taylor, PhD, Spaulding Rehabilitation Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: 2024P003589
Record Dates: First submitted 2025-02-07; First posted 2025-02-14 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Healthy
Keywords: Q-Collar; Cerebrovascular Blood Flow Regulation; Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: The study will involve two identical study sessions at Spaulding Hospital Cambridge performed with or without the participant wearing a properly fitted Q-Collar. Both study sessions will be completed in a 4-week period, with the order of study sessions assigned randomly during the consent procedure. All studies will be performed between 8AM-1PM in the Cardiovascular Research Laboratory. Participants will be NPO for two hours, will have refrained from caffeine consumption for 24 hours, and from vigorous physical activity for 48 hours prior to study start time. Participants will have refrained from all medications and nutraceuticals for 48 hours prior to study. Women will be asked to provide a urine sample to determine that they are not pregnant. Upon arrival, subjects will be given 5 ml water per kg body mass to minimize potential effects of hydration status.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Cerebrovascular Control with Q-Collar (Experimental): Participants will undergo measurements of cerebral blood flow during changes in body position (sit-to-stand) and resistance breathing tasks while wearing a properly fitted Q-collar to evaluate how the Q-Collar affects cerebrovascular responses to rapid and sinusoidal shifts in blood pressure.
  Interventions: Device: Q30 Q-Collar
- Cerebrovascular Control without Q-Collar (Placebo Comparator): Participants will undergo measurements of cerebral blood flow during changes in body position (sit-to-stand) and resistance breathing tasks without wearing a Q-collar.
  Interventions: Other: Not wearing Q-Collar

INTERVENTIONS:
Device: Q30 Q-Collar — Participants will complete a series of tests (sit-to-stand, resistive breathing, and graded bike test) while wearing a Q-Collar.
  Other Names: Q-Collar
  Arms: Cerebrovascular Control with Q-Collar
Other: Not wearing Q-Collar — Participants will undergo the same study procedures without wearing the Q-Collar.
  Arms: Cerebrovascular Control without Q-Collar

SUMMARY:
The goal of this clinical trial is to learn how the FDA-cleared Q-Collar device affects brain blood flow regulation during rest and exercise in healthy adults. The main questions this study aims to answer are:

1. How does the Q-Collar affect brain blood flow when there are quick changes in blood pressure, like when standing up quickly, or when breathing against resistance?
2. How does the Q-Collar affect brain blood flow during exercise?

Researchers will compare sessions where participants wear the Q-Collar to sessions where they do not wear the device to see if the Q-Collar improves brain blood flow during both rest and exercise.

Participants will:

* Complete two study visits, each 1 to 4 weeks apart.
* Perform a series of tasks, including standing tests, breathing tests, and exercise on a stationary bike, while their heart rate, brain blood flow, and other body functions are monitored.
* Wear the Q-Collar during one of the sessions and not wear it during the other session. The order of the sessions will be randomly assigned.

DETAILED DESCRIPTION:
We are doing this research to improve our understanding of how a FDA-cleared device, called the Q-Collar, affects brain blood flow regulation both at rest and in response to exercise. Participants will be asked to complete two study visits over a period of 1 to 4 weeks. Each visit will involve identical assessments, with the Q-Collar worn during one session and not during the other. The order of the sessions will be randomly assigned.

Each visit consists of three main tasks:

Standing Test (approximately 10 minutes): Participants will perform a series of movements, standing up from a seated position, while heart rate, breathing, and brain function are monitored. This test will be repeated three times per session.

Resistive Breathing Test (approximately 10 minutes): Using a mouthpiece that controls breathing difficulty, participants will breathe at specific depths and rates while sensors track gases, heart, lung, and brain activity. This task will be completed once per session.

Stationary Biking Exercise Test (approximately 30 minutes): Participants will perform an exercise test on a stationary bike while monitors measure heart rate, breathing gases, blood pressure, and brain blood flow. The test begins with a 2-minute warm-up, followed by progressively more challenging pedaling, with resistance adjusted based on body weight. Difficulty increases every 1 to 2 minutes until the required pace can no longer be maintained. Periodic ratings of exertion will be recorded. The session concludes with a 2-minute cool-down after maximum effort is reached.

ELIGIBILITY:
Inclusion Criteria:

* healthy individuals between the ages of 18 to 30 years old

Exclusion Criteria:

* History of concussion or other brain injury resulting in loss or alteration in consciousness or other change in cognition within 24 months of study visit
* High cardiac risk according to the American College of Sports Medicine (ACSM)11
* Ongoing active treatment with a cardioactive drug
* Inability to stand from a seated position unassisted
* History of a neurologic disorder or neurosurgery intervention
* Pregnancy
* Any current, serious, chronic medical or psychiatric disease that in the Principal Investigator's or co-investigator's judgment may interfere with study participation or data integrity
* Unable or unwilling to provide informed consent

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07-23 (Actual); Primary Completion 2026-07-23 (Estimated); Study Completion 2026-08-23 (Estimated)

PRIMARY OUTCOMES:
Sit-to-Stand Test: Autoregulatory Slope | 2 study visits within a 4 week time frame
  The slope of the autoregulatory curve, representing the change in cerebral blood flow in response to rapid shifts in blood pressure during the sit-to-stand transition.
Resistance Breathing Test: Autoregulatory Gain | 2 study visits within a 4 week time frame
  The autoregulatory gain, which reflects the brain's ability to maintain stable cerebral blood flow during sinusoidal fluctuations in blood pressure induced by resistance breathing.
Graded Bike Test: Change in Cerebral Blood Flow | 2 study visits within a 4 week time frame
  The change in cerebral blood flow velocity (CBFV) during the graded exercise test, assessed by Transcranial Doppler ultrasonography, indicating how cerebral blood flow responds to increasing physical exertion.

CONTACTS AND LOCATIONS:
Overall Officials: J. Andrew Taylor, MS, PhD, Principal Investigator — Harvard Medical School/Spaulding Rehabilitation Hospital
Locations (1):
- Spaulding Rehabilitation Hospital, Cambridge, Massachusetts, United States